CLINICAL TRIAL: NCT02779387
Title: Efficacy of Laparoscopic Surgery Combined With GnRH-a in the Treatment of Endometriosis Associated Infertility: A Multicenter, Prospective, Randomized-control-trial
Brief Title: Reproductive Outcome of EM Treated by GnRH-a Associated With Laparoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yu xiaoming, Clinician from Department of reproductive medicine.Secretary general of Fallopian tube group,Society for reproductive surgery, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU01001
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Infertility Associated With Endometriosis
Keywords: GnRH-a; endometriosis; efficiency
MeSH Terms: conditions — Endometriosis | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GnRH-a (Experimental): patients treated with GnRH-a after surgery and Outpatient guidance
  .
  Interventions: Drug: Goserelin Acetate
- non GnRH-a (No Intervention): patients treated with outpatient guidance only.

INTERVENTIONS:
Drug: Goserelin Acetate
  Arms: GnRH-a

SUMMARY:
This study is a multicenter, randomized-control-trial. This study select 1184 Infertile patients associated with endometriosis diagnosed by laparoscopy surgery. Patients are going to be divided into two groups according to 1:1 ratio randomly assigned to receive GnRH-a. Cumulative pregnancy rate, end of treatment to natural pregnancy time, accept the assisted reproductive treatment rate, miscarriage rate, live birth rate will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients
* Endometriosis I-II phase：according to Revised American Society for Reproductive Medicine classification of endometriosis: 1996
* BMI:19-28 kg/㎡
* Ovarian reserve function is normal（M2-5：bilateral antral follicles≥6 FSH：5-12U/ml）

Exclusion Criteria:

* Male factor causes infertility
* hydrosalpinx or salpingemphraxis
* Uterine malformation
* Uterine cavity lesion
* Contra-indications for GnRH-a
* not willing to participate

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1184 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Cumulative pregnancy rate | 18 month after surgery
  Cumulative pregnancy rate of 18 month after surgery
Time interval between surgery and natural pregnancy | 18 month after surgery
  Time interval between surgery and natural pregnancy
miscarriage rate | 18 month after surgery
  miscarriage rate of patients who get natural pregnancy

IPD SHARING:
Plan to Share IPD: Yes
Willing to share IPD